CLINICAL TRIAL: NCT01001871
Title: Seasonal Impact of Iron Fortification on Malaria Incidence in Ghanaian Children
Brief Title: Treatment of Iron Deficiency Anemia in Malaria Endemic Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000013476
Record Dates: First submitted 2009-10-21; First posted 2009-10-27 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: Iron deficiency anemia; Sprinkles®; micronutrients; malaria incidence; iron supplement
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Vitamins; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin/mineral fortificant with iron (Experimental)
  Interventions: Dietary Supplement: Sprinkles®
- Vitamin/mineral fortificant without iron (Placebo Comparator)
  Interventions: Dietary Supplement: vitamin/mineral fortificant without iron

INTERVENTIONS:
Dietary Supplement: Sprinkles® — powdered vitamin/mineral fortificant WITH iron sprinkled onto food once a day for 5 months
  Arms: Vitamin/mineral fortificant with iron
Dietary Supplement: vitamin/mineral fortificant without iron — powdered vitamin/mineral fortificant WITHOUT iron sprinkled onto food once a day for 5 months
  Arms: Vitamin/mineral fortificant without iron

SUMMARY:
Iron deficiency and iron deficiency anemia (IDA) are the most prevalent micronutrient deficiencies on a worldwide basis, especially in developing countries. The impact of severe IDA can have mortal consequences, since without adequate hemoglobin, the brain and body become deprived of oxygen and, if allowed to continue, death may ensue. It has been shown that iron supplementation in infants and young children can enhance child development, however, it may also result in increased rates of malaria in high burden areas.

The primary objective of this study is to determine the impact of providing encapsulated iron (as a powder added to complementary foods) on the susceptibility to clinical malaria among anemic and non-anemic infants and young children (6-24 months of age) living in a high malaria burden area.

The value of performing this research in Ghana is primarily that malaria and anemia remain the most important causes of death and morbidity.

DETAILED DESCRIPTION:
Study Design:

The proposed study is a community-based blinded randomized controlled trial with 2 study arms that will be conducted in two phases:

* Phase I will take place during the dry season (December to April), when malaria transmission rates are lower. Eligible subjects (one per household) will be individually randomized to receive a daily dose of either a powdered vitamin/mineral fortificant containing 12.5 mg of iron (plus ascorbic acid, vitamin A and zinc), or a placebo (containing all micronutrients excluding iron), added to complementary foods, for 5 months.
* Phase II will take place during the wet season (June to October), when malaria transmission rates are higher. Eligible subjects, who did not participate in Phase I, will be individually randomized to one of the two study arms as described above and followed for 5 months.

A dual phase design, with two unique cohorts, was chosen so that preliminary results (at the end of phase 1) could be assessed by an independent Data Safety and Monitoring Committee. It is possible that during the dry season no impact of iron will be detected, while during the wet season, an impact will be observed. With this possible outcome, it is potentially feasible to translate this knowledge into a Ministry of Health Program to only provide iron supplementation (fortification) during the dry months of the year (December to April).

ELIGIBILITY:
Inclusion Criteria:

* Age 6-24 months
* Ingesting weaning food in addition to breastmilk
* Free from malaria or other major illnesses
* Afebrile
* Living in Brong Ahafo Region of Ghana for duration of intervention and follow-up

Exclusion Criteria:

* Severe anemia (hemoglobin <70g/L)
* Weight-for-height <-3 z-score(severe wasting)
* Kwashiorkor (defined as evidence of edema)
* Congenital abnormality
* Treatment with iron supplements within the past 6 months
* Presence of any chronic illness

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3880 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
incidence of clinical malaria (if fever recorded a blood sample will be taken to determine parasite species and count) | 5 months

SECONDARY OUTCOMES:
changes in anemia status (blood levels of: haemoglobin(Hb) , ferritin (SF)) | 5 months
severity of clinical malaria (blood parasite count) | 5 months
cerebral malaria (defined by a parasite count >5000/μL blood and a concurrent score of <2 on the Blantyre coma scale, with or without convulsions) | 5 months
hospitalization (documentation of hospitalization for any reason) | 5 months
death | 5 months
pneumonia (defined by the presence of a cough or breathing difficulties, tachypnea, lower chest wall indrawing, and the appearance of consolidation or pleural effusion on a chest X-ray) | 5 months
diarrhea (defined by >3 loose or watery stools in the previous 24 hours) | 5 months
dehydration (defined by lethargy, sunken eyes, and decreased skin turgor [>2 seconds for skin to return following a skin pinch]) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Zlotkin, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- Kintampo Health Research Centre, Kintampo, Ghana

REFERENCES:
- [Derived] Tchum SK, Sakyi SA, Arthur F, Adu B, Abubakar LA, Oppong FB, Dzabeng F, Amoani B, Gyan T, Asante KP. Effect of iron fortification on anaemia and risk of malaria among Ghanaian pre-school children with haemoglobinopathies and different ABO blood groups. BMC Nutr. 2023 Mar 23;9(1):56. doi: 10.1186/s40795-023-00709-w. PMID 36959634
- [Derived] Tchum SK, Sakyi SA, Adu B, Arthur F, Oppong FB, Dzabeng F, Amoani B, Gyan T, Poku-Asante K. Impact of IgG response to malaria-specific antigens and immunity against malaria in pre-school children in Ghana. A cluster randomized, placebo-controlled trial. PLoS One. 2021 Jul 20;16(7):e0253544. doi: 10.1371/journal.pone.0253544. eCollection 2021. PMID 34283841
- [Derived] Aimone AM, Brown P, Owusu-Agyei S, Zlotkin SH, Cole DC. Impact of iron fortification on the geospatial patterns of malaria and non-malaria infection risk among young children: a secondary spatial analysis of clinical trial data from Ghana. BMJ Open. 2017 Jun 6;7(5):e013192. doi: 10.1136/bmjopen-2016-013192. PMID 28592572
- [Derived] Aimone AM, Brown PE, Zlotkin SH, Cole DC, Owusu-Agyei S. Geo-spatial factors associated with infection risk among young children in rural Ghana: a secondary spatial analysis. Malar J. 2016 Jul 8;15:349. doi: 10.1186/s12936-016-1388-1. PMID 27391972
- [Derived] Zlotkin S, Newton S, Aimone AM, Azindow I, Amenga-Etego S, Tchum K, Mahama E, Thorpe KE, Owusu-Agyei S. Effect of iron fortification on malaria incidence in infants and young children in Ghana: a randomized trial. JAMA. 2013 Sep 4;310(9):938-47. doi: 10.1001/jama.2013.277129. PMID 24002280